CLINICAL TRIAL: NCT04421040
Title: Long-term Monitoring of Patients With Cardiac Amyloidosis With Implantable Event Monitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Omar Abou Ezzeddine, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-006298
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: TTR Cardiac Amyloidosis

STUDY DESIGN:
Intervention Model Description: Patients with TTR-wt cardiac amyloidosis will be monitored with an implantable loop recorder to determine frequency of atrial and ventricular arrhythmias. After 6 months the device will be explanted unless required for further clinical monitoring.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Biomonitor 3 (Experimental): Placement of Biotronik Biomonitor 3 Device for a 6 month period. After the 6 month monitoring period, the patient will have the Biotronik Biomonitor 3 device removed.
  Interventions: Device: Biotronik Biomonitor 3 implant of device; Device: Biotronik Biomonitor 3 explant of device

INTERVENTIONS:
Device: Biotronik Biomonitor 3 implant of device — The Biotronik Biomonitor 3 device will be implanted by the research team physician.
Device: Biotronik Biomonitor 3 explant of device — The Biotronik Biomonitor 3 device will be removed from the patient by the research team physician.

SUMMARY:
Researchers are gathering information to see if using an FDA approved implantable device can help with monitoring of your heart arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac biopsy or technetium pyrophosphate scintigraphy confirmed patients
* Stage I, II, and early and late stage III in numbers as described , irrespective of EF or NYHA functional class
* Patients aged 18 -85, both genders and of all races and ethnicities.
* Patients must be competent to give informed consent.
* Patients must be able to have the Biomonitor 3 implanted.
* Amyloid stage I-III patients with existing implantable cardiac devices such as pacemakers or defibrillators

Exclusion Criteria:

* Significant coronary artery disease > 75% luminal stenosis in at least 1 epicardial vessel (by cardiac catheterization or coronary computed tomography), or history of myocardial infarction or coronary revascularization.
* Congenital heart disease.
* Pregnant patients
* Patients whose heart failure is felt to be secondary to primary valvular disease (>moderate/severe mitral regurgitation), uncorrected thyroid disease, obstructive or hypertrophic cardiomyopathy, pericardial disease or a systemic illness.
* Absolute contraindications to cardiac MRI (such as renal failure with GFR<30%).
* Unwilling or unable to provide informed consent.
* Patients with other life threatening diseases that would likely decrease their life expectancy over the next four years.
* Patients who are post cardiac transplant.
* Difficulty to attend the follow-up schedule due to a history of medical noncompliance, difficulty, or unwillingness to return to the study center for follow up.
* Evidence of ongoing bacteremia or sepsis preventing implantation of a device
* Unwilling or able to have the Biomonitor 3 interrogated

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Abou Ezzeddine, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biomonitor 3
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Biomonitor 3
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Sudden Death
Description: Total number of patients to experience sudden death
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Biomonitor 3
Number analyzed (Participants) | 24
Participants | 0

2. Primary Outcome: Atrial Arrhythmias
Description: Total number of participants to experience atrial arrhythmias
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Biomonitor 3
Number analyzed (Participants) | 24
Participants | 10

3. Primary Outcome: High Grade Atrioventricular (AV) Block
Description: Total number of patients with high grade atrioventricular (AV) block.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Biomonitor 3
Number analyzed (Participants) | 24
Participants | 2

4. Primary Outcome: Permanent Pacemaker Implantation
Description: Total number of patients requiring permanent pacemaker implantation.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Biomonitor 3
Number analyzed (Participants) | 24
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant for 6 months, from baseline until device ex-plantation.
Arm/Group | Biomonitor 3
All-Cause Mortality (participants affected / at risk) | 2/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 8/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biomonitor 3 (N=24)
Heart palpitations (Cardiac disorders) | 4 (4)
Fatigue (General disorders) | 3 (3)
Syncope (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT04421040/Prot_SAP_000.pdf